CLINICAL TRIAL: NCT01817777
Title: A Pharmacy Based Open Study to Evaluate Whether Pack Size Affects Compliance for Subjects Diagnosed With Diabetes Type II Who Are Established on Metformin Treatment
Brief Title: An Open Study to Evaluate Whether Pack Size Affects Compliance of Metformin Treatment in Subjects With Type II Diabetes
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: It's no longer feasible to continue to recruit patients into the study as severe recruitment difficulties have been experienced since the study start
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 116086
Record Dates: First submitted 2013-03-21; First posted 2013-03-25 (Estimated); Results first posted 2014-09-30 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Socioeconomic category; Medication compliance; Metformin; small pack
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin Small Pack Arm (Experimental): All subjects in the study will be initially followed for an 8-week observational phase during which subjects will visit the pharmacy and purchase metformin following their usual routines. After 8-weeks subjects will be randomised to one of the 2 treatments arms. Subjects in the metformin small pack arm will receive medication free of charge in a small pack. Dosing of metformin will not be dictated by the protocol. Subjects will remain on their prescribed dose of metformin throughout the study, unless a change is recommended by their physician.
  Interventions: Drug: Metformin Small Pack
- Metformin Large Pack Arm (Experimental): All subjects in the study will be initially followed for an 8-week observational phase during which subjects will visit the pharmacy and purchase metformin following their usual routines. After 8-weeks subjects will be randomised to one of the 2 treatments arms. Subjects in the metformin large pack arm will receive medication free of charge in a large, monthly pack. Dosing of metformin will not be dictated by the protocol. Subjects will remain on their prescribed dose of metformin throughout the study, unless a change is recommended by their physician.
  Interventions: Drug: Metformin Large Pack

INTERVENTIONS:
Drug: Metformin Small Pack — A single small pack of metformin will consist of a blister package containing 10 pills with a patient information leaflet in local language. The small packs will be available at each site in the following doses: 500 mg, 850 mg, and 1000 mg. The small pack size of metformin is not yet marketed. Small pack metformin will be provided by GSK as GSK brand metformin.
  Arms: Metformin Small Pack Arm
Drug: Metformin Large Pack — The large pack will consist of 1 month's supply of metformin.
  Arms: Metformin Large Pack Arm

SUMMARY:
MTF116086 is an open-label, randomised, parallel-design study in subjects with type II diabetes. The study is site-based, with local pharmacies serving as the sites and pharmacists as principal investigators for the sites. All subjects will enter an initial 8-week observational phase during which purchase behaviour and compliance with usual metformin use will be observed and recorded. At the end of the observational phase, subjects will be randomised to one of the two arms (metformin small pack vs. metformin large pack) for a 20-week interventional phase. The medication in the interventional phase is provided to the subjects free of charge. HbA1c will be collected for all subjects during Week 0, Week 8, and Week 28. Subjects will be asked questions about their tablet compliance, their satisfaction with the pack size they received and reasons for missing doses throughout the interventional phase by the pharmacist. The pharmacy visit on Week 28 will be end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of age >=18 years
* Diagnosis of type II diabetes
* HbA1c value no higher than 9.0%
* Evidence of physician-supplied prescription for metformin use
* Stable dose of metformin for 3 months prior to enrolment
* Written informed consent from the subject

Exclusion Criteria:

* Current use of any anti-diabetic medication other than metformin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-05; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Argentina (5):
  - GSK Investigational Site, Correintes
  - GSK Investigational Site, Corrientes
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, Provincia de Buenos Aires
  - GSK Investigational Site, San Miguel de Tucumán

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 116086 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116086 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116086 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116086 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116086 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116086 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116086 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants aged >=18 years with a diagnosis of Type II diabetes mellitus (T2DM) and a glycated hemoglobin (HbA1c) value no higher than 9.0%; with evidence of a physician-supplied prescription for metformin use and on a stable dose of metformin for 3 months prior to enrollment; and on no anti-diabetic medication other than metformin were enrolled.
Pre-assignment Details: Enrolled participants entered an 8-week Observational Phase (OP) prior to randomization to one of the treatment arms, followed by a 20-week Interventional Phase (IP). A total of 288 participants were planned; however, the study was prematurely discontinued when 36 participants had entered the OP. Of these 36, 31 had entered the IP.
Groups:
- Routine Metformin: Participants were followed during an 8-week Observational Phase. During this phase, participants visited the pharmacy and purchased metformin (MTF) as per their usual routines.
- Small Pack Metformin: Each participant received a small pack of MTF for an individualized dose depending on their diabetes treatment needs. The small packs were available at each site in the following doses of MTF: 500 milligrams (mg), 850 mg, and 1000 mg. Participants on MTF twice daily received one small pack at each visit (sufficient for 5 days of treatment). Participants on MTF three times daily received two small packs at each visit (sufficient for 6 days of treatment).
- Large Pack Metformin: Each participant received a large pack of MTF for an individualized dose depending on their diabetes treatment needs. The large pack consisted of one month's supply of metformin.
Period: Observational Phase (8 Weeks)
Arm/Group | Routine Metformin | Small Pack Metformin | Large Pack Metformin
Started | 36 | 0 | 0
Completed | 31 | 0 | 0
Not Completed | 5 | 0 | 0
Not completed — Lost to Follow-up | 3 | 0 | 0
Not completed — Early Study Termination | 2 | 0 | 0
Period: Interventional Phase (20 Weeks)
Arm/Group | Routine Metformin | Small Pack Metformin | Large Pack Metformin
Started | 0 | 16 | 15
Completed | 0 | 11 | 10
Not Completed | 0 | 5 | 5
Not completed — Withdrawal by Subject | 0 | 3 | 0
Not completed — Lost to Follow-up | 0 | 1 | 2
Not completed — Early Study Termination | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Small Pack Metformin | Large Pack Metformin | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.3 (12.01) | 56.3 (10.52) | 57.3 (11.17)
Gender [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 9 | 8 | 17
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasic (White) | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c Values at Week 28
Description: HbA1c was tested with a point-of-care device, which required a finger prick to obtain blood and provided an immediate result upon analysis in the device. HbA1c was tested at pharmacy visits corresponding to three time points: enrollment (Week 0), Baseline (Week 8), and End of Study (Week 28). The difference in the mean change from Baseline was to be calculated between the treatment arms (small pack minus large pack), and the 2-sided 95% confidence interval for the difference in mean change in HbA1c was to be calculated. However, because the study was terminated early, and the sample size was reduced, the statistical hypotheses defined in the protocol were not tested due to insufficient power. Therefore, the final analyses were limited to descriptive statistics. The percentage HbA1c is a measure of how much of the hemoglobin in the blood has become glycated (chemically bounded to glucose).
Time Frame: Baseline (Week 8) and Week 28
Population: Per Protocol Population: all participants in the Intent-to-Treat Population (randomly assigned to treatment and who received >= 1 dose [or any portion of a dose] of study medication and had an HbA1c test at Week 8) who did not have a protocol violation
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Small Pack Metformin | Large Pack Metformin
Number analyzed (Participants) | 8 | 9
Percentage | -0.026 (0.5511) | -0.109 (0.8631)

2. Secondary Outcome: Mean Percent Compliance Throughout the Interventional Phase
Description: Compliance for the study was estimated as a percentage, with the denominator defined as the number of pills dispensed by the pharmacist and the numerator defined as the number of pills taken, accounting for remaining pills at subsequent pharmacy visits.
Time Frame: From Randomization to Week 28
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: Percent compliance
Arm/Group | Small Pack Metformin | Large Pack Metformin
Number analyzed (Participants) | 8 | 9
Percent compliance | 74.08 (11.439) | 90.83 (4.778)

3. Secondary Outcome: Mean Percent Compliance Throughout the Observational Phase, Per Treatment They Were Randomized to in the Interventional Phase
Description: Compliance was estimated during the 8-week Observational Phase for usual metformin treatment. During the Observational Phase, compliance was measured by monitoring the number of pill dispensed and the return of the pills or tablets.
Time Frame: From enrollment to Week 8
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: Percent compliance
Arm/Group | Small Pack Metformin | Large Pack Metformin
Number analyzed (Participants) | 8 | 9
Percent compliance | 65.61 (13.901) | 88.07 (22.303)

4. Secondary Outcome: Number of Participants Who Took Zero Metformin Pills for the Indicated Number of Days
Description: The number of days on which no metformin pills were taken by participants was summarized.
Time Frame: Week 28
Population: Per Protocol Population
Measure: Number; unit: Participants
Arm/Group | Small Pack Metformin | Large Pack Metformin
Number analyzed (Participants) | 8 | 9
Participants
  1 day | 2 | 1
  2 days | 1 | 1
  3 days | 0 | 0
  4 days | 0 | 0
  5 days | 0 | 1
  6 days | 0 | 0
  7 or more days | 4 | 2

5. Secondary Outcome: Number of Participants With Diabetes Disease Management Modifications
Description: Throughout the duration of the study, participants remained on their recommended metformin dosing regimens, unless a change in metformin dose was prescribed by their physician. The number of participants who received additional diabetes therapy for the management of diabetes was summarized.
Time Frame: Week 28
Population: Per Protocol Population
Measure: Number; unit: Participants
Arm/Group | Small Pack Metformin | Large Pack Metformin
Number analyzed (Participants) | 8 | 9
Participants | 0 | 1

6. Secondary Outcome: Number of Participants Who Required a Non-routine Health Care Professional Visit for Diabetes
Description: The number of participants who visited a health care professional for diabetes management during the study was summarized.
Time Frame: Week 28
Population: Per Protocol Population
Measure: Number; unit: Participants
Arm/Group | Small Pack Metformin | Large Pack Metformin
Number analyzed (Participants) | 8 | 9
Participants | 5 | 6

7. Secondary Outcome: Number of Participants Who Preferred Their Treatment Regimens (Interventional Arm Treatment [Large or Small Pack Metformin]) to How They Previously Took Their Medication
Description: Number of participants who preferred their treatment regimens (interventional arm treatment [large or small pack metformin]) to how they previously took their medication are presented.
Time Frame: Week 28
Population: Per Protocol Population
Measure: Number; unit: Participants
Arm/Group | Small Pack Metformin | Large Pack Metformin
Number analyzed (Participants) | 8 | 9
Participants | 8 | 8

8. Secondary Outcome: Number of Participants Who Missed Metformin Days/Doses for the Indicated Reasons
Description: The number of particiapnts who missed days or doses of metformin was summarized.
Time Frame: Week 28
Population: Per Protocol Population
Measure: Number; unit: Participants
Arm/Group | Small Pack Metformin | Large Pack Metformin
Number analyzed (Participants) | 8 | 9
Participants
  Lost Medication | 0 | 0
  Forgetful | 3 | 5
  Other | 3 | 1

9. Secondary Outcome: Number of Participants Withdrawn From the Study Due to the Following Reasons: Withdrawal of Informed Consent; Lost to Follow-up
Description: The number of participants who voluntarily discontinued participation in the study at any time or who were withdrawn by the investigator for pre-defined reasons was summarized.
Time Frame: Week 28
Population: Observational Population: all participants enrolled into the study. If an enrolled participant withdrew from the study prior to the Week 8 visit, all available data on the participant was included in the Observational Population.
Measure: Number; unit: Participants
Arm/Group | Small Pack Metformin | Large Pack Metformin
Number analyzed (Participants) | 16 | 15
Participants | 4 | 2

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of interventional study treatment (Week 8) until Week 28.
Description: SAEs and non-serious AEs were collected in members of the Safety Population, comprised of all participants who received >=1 dose of study medication. Data were analyzed according to the actual treatment the participant received.
Arm/Group | Small Pack Metformin | Large Pack Metformin
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 5/16 | 2/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Small Pack Metformin (N=16) | Large Pack Metformin (N=14)
Dizziness (Nervous system disorders) | 1 | 0
Cold (Infections and infestations) | 2 | 0
Cataract (Eye disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Endocervical polyp (Reproductive system and breast disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.